CLINICAL TRIAL: NCT06497842
Title: The Effect of Perceived Effort in Resistance Training on Glycemic Control and Psychological Responses in Individuals Living With Type 2 Diabetes Mellitus: a Randomized-controlled, Parallel Group, Clinical Trial
Brief Title: Effort During Resistance Training in Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRRC#24-101
Record Dates: First submitted 2024-06-28; First posted 2024-07-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Resistance training; Degree of effort; Glycemic control; Continuous glucose monitoring

STUDY DESIGN:
Intervention Model Description: Participants will undergo anthropometrics, familiarization, and strength test, and will be randomized to a high-effort, or a low-effort resistance training protocol, that will be carried out 2 days/week, for 16 weeks, and will be composed of 7 exercises (hex bar squat, seated chest press, leg press, lat pulldown, leg extension, shoulder press, leg curl, always in this order). Load will be set at 10-RM load (75% 1-RM). Participants will be instructed to perform the concentric (lifting) phase of the repetition as fast as they can (~0.5 seconds), and to perform the eccentric phase in 2 seconds. Psychological responses (perceived exertion, enjoyment, feeling scale, discomfort, and self-efficacy) will be assessed. Anthropometrics will be repeated after training, and before and after the training period, glycemic control will be assessed via a continuous glucose monitoring device. The main outcomes will be compared between training interventions, pre-training data will used as comparator.
Who Masked: Outcomes Assessor
Masking Description: Data and statistical analysis will be performed by a researcher blinded to groups and participants' identities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-effort (Experimental): The high-effort protocol will entail performing 3 sets per exercise, 8 repetitions per set, ~2.5 seconds per repetition, with 120 seconds between sets and exercises.
  Interventions: Behavioral: High-effort resistance exercise training
- Low-effort (Experimental): The low-effort protocol will entail performing 6 sets per exercise, 4 repetitions per set, ~2.5 seconds per repetition, with 60 seconds between sets and exercises.
  Interventions: Behavioral: Low-effort resistance exercise training

INTERVENTIONS:
Behavioral: High-effort resistance exercise training — Six sets per exercise, 8 repetitions per set.
  Arms: High-effort
Behavioral: Low-effort resistance exercise training — Three sets per exercise, 4 repetitions per set.
  Arms: Low-effort

SUMMARY:
In this study the primary aims are to investigate the effect of resistance exercise training with different degrees of effort on glycemic control and psychological variables in individuals living with type 2 diabetes mellitus. As a secondary aim, investigate adherence and dropout rates and reasons for dropping out and adhering or not to the protocols.

DETAILED DESCRIPTION:
Resistance exercise training can be both effective for the management of type 2 diabetes mellitus (T2DM) and appealing for individuals living with T2DM, and has been shown to be a viable exercise prescription option for this population. It has been suggested that the degree of effort is important for acute improvements in glucose metabolism and insulin sensitivity in individuals living with T2DM, although direct evidence of that is lacking. However, performing resistance exercise sets with a high degree of effort is associated with higher perceived exertion and discomfort, increased muscle soreness, negative perceptual responses, and higher neuromuscular fatigue and muscle damage. Taken together, these negative perceptual and physiological responses to resistance exercise sets performed with high degree of effort might negatively affect enjoyment, self-efficacy, and motivation during a resistance exercise session, ultimately reducing long-term adherence.

The primary aim of this study is to assess the effects resistance exercise training with different degrees of effort on glycemic control and psychological responses in individuals living with T2DM. Also, perceptual responses will be assessed to investigate how feelings experienced during resistance exercise training are altered relative to different degrees of effort. The hypothesis is that glycemic control will not be affected by the degree of effort, and improvements will be observed regardless of that. Also, it is hypothesized that the degree of effort will be associated with better psychological responses. The secondary aim of this study is to investigate and report adherence rate and reasons for adhering or not to the protocols. It is anticipated that adherence will be associated with the degree of effort and psychological responses experienced during training.

ELIGIBILITY:
Inclusion Criteria:

* Living with type 2 diabetes mellitus

Exclusion Criteria:

* Have a significant cognitive impairment,
* Are non-ambulatory,
* Have lower extremity amputation,
* Have renal failure,
* Have liver disease,
* Have uncontrolled hypertension (>160 mmHg systolic and/or >100 mmHg diastolic),
* Have unstable cardiovascular disease,
* Have a history of severe cardiovascular problems,
* Have decompensated heart failure,
* Have uncontrolled arrhythmias,
* Have severe pulmonary hypertension (mean pulmonary arterial pressure >55 mm Hg),
* Have severe and symptomatic aortic stenosis,
* Have acute myocarditis, endocarditis, or pericarditis,
* Have aortic dissection,
* Have Marfan syndrome,
* Have unrepaired aortic aneurysm,
* Have proliferative diabetic retinopathy,
* Have rapidly progressive terminal illness,
* Are unable to perform resistance exercise to due preexisting musculoskeletal conditions (e.g., joint pain, chronic injury or tendinopathy),
* Are under biguanide (metformin) treatment, but are taking for less than 3 months,
* Have taken drugs known to increase the risk of tendon disorders (e.g., tendinopathy and tendon rupture) within the last 6 months. These drugs include, but may not be limited to: fluoroquinolones, glucocorticoids, aromatase inhibitors, anabolic steroids, antiretrovirals, isotretinoin, cephalexin, rituximab, sitagliptin, cephalosporins, azithromycin, and sulfonamides.
* Are pregnant or trying to become pregnant during the study,
* Are prisoners,
* Are persons that require a legally authorized representative.

Temporary exclusions include:

* Being subjected to recent surgeries for which resistance training is not recommended,
* Have symptomatic hernias,
* Have acute illness,
* Have recent fractures, or other injuries until resolved.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Glucose concentration | For 60 hours before the first training session and for 60 hours after the last (32nd) training session
  Average glucose concentration (measured in milligrams per deciliter of blood, with a continuous glucose monitoring device)

SECONDARY OUTCOMES:
Adherence to the resistance training protocols | From date of randomization until the date of first documented dropout from any cause, assessed up to 16 weeks (the end of the training period)
  Adherence rate assessed using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Flavio De Castro Magalhaes, PhD, Principal Investigator — Assistant Professor
Locations (1):
- UNM Exercise Physiology Lab, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
For sharing the data generated the Open Science Framework (OSF) platform will be used. Before data sharing, all personal identifiers will be stripped from the data. Specifically, any direct identifiers (e.g., name, email addresses, phone and cell phone numbers), date identifiers (e.g., birthday, date of disease diagnosis, dates patients participated in data collection), location identifiers (e.g., personal or professional addresses, zip codes), links to external datasets identifiers (e.g., social media accounts) will be removed. Furthermore, participants will be represented by an identification string generated randomly (www.random.org/strings/), and their data will be inserted in the files in a random order, not associated with the order they were enrolled. Thus, data will be entirely de-identified before sharing, in order to protect sensitive personal information and privacy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The anticipated date for data sharing will be 6 months after publication of data or 18 months after award end date, whatever happens first.
Access Criteria: Open access

DOCUMENTS (1):
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT06497842/ICF_000.pdf